CLINICAL TRIAL: NCT05800353
Title: Nd:YAG Laser Vitreolysis for Symptomatic Vitreous Floaters
Acronym: VVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dongyang People's Hospital (Other)
Responsible Party: Principal Investigator, Zhou Hangshuai, Deputy chief physician of ophthalmology, Dongyang People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DongyangPH
Record Dates: First submitted 2023-03-10; First posted 2023-04-05 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Weiss Ring
Keywords: Vitreous floaters; vitreolysis; Nd:YAG laser
MeSH Terms: conditions — vitreous floaters

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- early treatment group (Experimental): Participants in the early treatment group will receive a YAG laser vitreolysis immediately and a sham laser treatment three months later.
  Interventions: Procedure: YAG vitreolysis
- delayed treatment group (Experimental): Participants in the delayed treatment group will receive a sham laser treatment immediately and a YAG laser vitreolysis three months late.
  Interventions: Procedure: YAG vitreolysis

INTERVENTIONS:
Procedure: YAG vitreolysis — A Karickoff lens with goniosol will be used to perform the YAG vitreolysis. The number of shots will be determined at the discretion of the treating physician. A focus offset may be used at investigator discretion. Single shot mode will be used. The maximum energy per pulse will be 7 mJ. The endpoint of treatment is the vaporization of the Weiss ring into gas, as well as the disruption of it into smaller fragments as well as any other vitreous opacities deemed visually significant by the treating physician.
  Sham laser treatment will be applied under the same procedure used for laser treatment but by turning the laser power down to 0.3 mJ and using a separate lens covered by a filter that absorbs the power, so no laser enters the eye.
  Other Names: Sham YAG vitreolysis

SUMMARY:
The goal of this clinical trial is to compare in the efficacy and safety of Nd:YAG laser vitreolysis for symptomatic vitreous floaters. The main question it aims to answer are:

• examine the efficacy and safety in treating early onset of vitreous floaters （Weiss ring） using Nd:YAG laser vitreolysis.

Participants with symptomatic floaters for one month will be randomly divided into two groups：early treatment group and delayed treatment group. Participants in the early treatment group will receive a YAG laser vitreolysis immediately and a sham laser treatment three months later, while participants in the delayed treatment group will receive a sham laser treatment immediately and a YAG laser vitreolysis three months late.

Researchers will compare the two groups to see the efficacy and safety of early YAG laser vitreolysis for symptomatic vitreous floaters.

ELIGIBILITY:
Inclusion Criteria:

1. Self-rating of visual disturbance by the floaters must be at least 4 on a 0-10 scale, with 0 being no symptoms to 10 being debilitating symptoms.
2. Symptomatic Weiss ring (PVD) must be at least 2mm away from the retina and 5 mm from the posterior lens capsule of the crystalline lens, as measured on B-scan. For pseudophakic patients, there is no minimum required distance from the intraocular lens.
3. Able to position for the YAG laser procedure.
4. Accept the risks of YAG laser including but not limited to retinal detachment, intraocular hemorrhage, retinal damage, cataract formation, optic nerve damage, inflammation, and irreversible loss of vision.
5. Willing and able to comply with clinic visits and study-related procedures
6. If the patient has two symptomatic eyes, only one eye can be randomized and included in the study.
7. Provide signed informed consent

Exclusion Criteria:

1. History of retinal tear, retinal detachment, or uveitis in the study eye
2. History of diabetic retinopathy, macular edema, retinal vein occlusion, or aphakia in the study eye
3. History of glaucoma or high intraocular pressure defined as having a history of glaucoma surgery or currently taking two or more topical glaucoma medications in the study eye

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Subjective improvement in floater symptoms | 3 Months
  Doctor/Surveyor: Hi there, have you experienced any visual disturbances such as floaters? On a scale of 0 to 10, with 0 meaning no symptoms and 10 meaning symptoms that significantly impact your daily life, how would you rate the severity of your visual disturbance caused by the floaters?
Visual Functioning Questionnaire-25 | 3 Months
  Mean change in the National Eye Institute Visual Functioning Questionnaire-25 (NEI VFQ-25). The Visual Functioning Questionnaire-25 (VFQ-25) is a self-reported questionnaire designed to measure a patient's visual function and its impact on their quality of life. The VFQ-25 consists of 25 items, which assess various domains of vision-related quality of life, such as general vision, near and distance activities, driving, social functioning, and mental health. The minimum value for the VFQ-25 is 0, which represents the worst possible visual function and quality of life, while the maximum value is 100, indicating the best possible visual function and quality of life. Higher scores on the VFQ-25 indicate a better outcome, indicating that the patient has better visual function and quality of life.

SECONDARY OUTCOMES:
Qualitative changes through OCT and fundus photography | 3 Months
  The objective evaluation of the improvement of vitreous floaters through OCT and fundus photography can be divided into five levels: worse, no change, mild improvement, significant improvement, and complete improvement.
Incidence and severity of ocular and systemic adverse events | 3 Months
  Incidence rates of retinal tears, retinal hemorrhage, retinal detachment, lens damage, and other related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Guangjin Zhao, Study Chair — Dongyang People's Hospital
Locations (1):
- Dongyang People's Hospital, Dongyang, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hangshuai Z, Yanhua J, Yao Z, Guangjin Z, Hongyan W, Fanlian C. Efficacy and safety of early YAG laser vitreolysis for symptomatic vitreous floaters: the study protocol for a randomized clinical trial. Trials. 2024 Jan 13;25(1):48. doi: 10.1186/s13063-024-07924-1. PMID 38218919